CLINICAL TRIAL: NCT00005230
Title: Epidemiology of Carotid Disease in Elderly Adults
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1110; R29HL039871 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Carotid Artery Diseases; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Carotid Artery Diseases; Atherosclerosis

SUMMARY:
To determine whether a population with isolated systolic hypertension (ISH) had a higher prevalence of carotid disease than a normotensive population matched for age and sex, and to determine specific risk factors for carotid disease.

DETAILED DESCRIPTION:
BACKGROUND:

The Systolic Hypertension in the Elderly Program was a multicenter controlled clinical trial supported by the NHLBI to study the cardiovascular and psychological effects of isolated systolic hypertension in the elderly and to determine the efficacy and evaluate possible adverse effects of drug treatment for this condition. A total of 4,736 patients were followed until 1991. Elderly individuals with isolated systolic hypertension are clearly at increased risk of both heart attack and stroke. This group has been shown in pilot studies to also have high prevalence of carotid disease and lower extremity arterial disease. Selected risk factors such as older age, male sex, and smoking were found to be related to an increased prevalence of disease. This study allowed validation of these initial observations.

DESIGN NARRATIVE:

This study was ancillary to the Systolic Hypertension in the Elderly Program (SHEP) clinical trial. Participants of the SHEP at the University of Pittsburgh were used for the hypertensive population. Patients screened for SHEP but rejected because of normal blood pressure were used for the controls. Carotid disease was assessed by duplex scanning, a noninvasive technique that combined real time B-mode ultrasound with Doppler ultrasound, producing a system capable of both vessel imaging and analysis of blood flow characteristics. Other evaluations included ankle systolic blood pressure measurements to detect lower extremity arterial disease, complete history and physical examination, electrocardiogram, blood lipoprotein levels, fasting insulin and glucose levels, hemoglobin, and hematocrit. Thus, the effects of various risk factors on the development of carotid atherosclerosis were evaluated as well as the relationship between carotid atherosclerosis and peripheral arterial disease of the lower extremities. The first six months of the study consisted of preparation and reproducibility testing of duplex scan measurements. During the following three years, duplex scans and other evaluations were completed on all 400 participants. During the final half of the fourth year, the first 100 duplex scans of hypertensive participants were repeated to determine whether it was possible to measure disease progression using this methodology. The study began in FY 1988 under R29HL39871 and continued in FY 1993 under R01HL50439.

The study was renewed in 1998 for an additional three years through June, 2003. The study continued to investigate the prevalence and prognostic value of subclinical atherosclerosis in the Pittsburgh SHEP cohort and a cohort of normotensive controls. Annual telephone follow-up of the remaining 178 SHEP participants and 168 controls continued. A final clinic visit included measures of coronary and aortic calcification using electron beam computed tomography (CT), pulse wave velocity as a measure of aortic stiffening and cognitive function testing. For the Pittsburgh SHEP cohort, the antihypertensive treatment effect was striking with event rates for the active and placebo groups continuing to diverge beyond the end of SHEP. Successful demonstration of a treatment effect on coronary calcium scores would be the first randomized data showing an antihypertensive effect directly in the coronary arteries. Risk factors for coronary calcification were evaluated, producing data of a type not yet available in the literature for older adults and not being collected in any other ongoing studies of the elderly. The added measures of vascular stiffness supplemented the extensive data on subclinical atherosclerosis already available for this cohort. The extent to which these measures predicted cardiovascular events was evaluated.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-07; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Tyrrell — University of Pittsburgh

REFERENCES:
- [Background] Sutton-Tyrrell K, Wolfson SK Jr, Thompson T, Kelsey SF. Measurement variability in duplex scan assessment of carotid atherosclerosis. Stroke. 1992 Feb;23(2):215-20. doi: 10.1161/01.str.23.2.215. PMID 1561650
- [Background] Sparrow D, O'Connor GT, Rosner B, Weiss ST. Methacholine airway responsiveness and 24-hour urine excretion of sodium and potassium. The Normative Aging Study. Am Rev Respir Dis. 1991 Sep;144(3 Pt 1):722-5. doi: 10.1164/ajrccm/144.3_Pt_1.722. PMID 1892316
- [Background] Sutton-Tyrrell K, Alcorn HG, Herzog H, Kelsey SF, Kuller LH. Morbidity, mortality, and antihypertensive treatment effects by extent of atherosclerosis in older adults with isolated systolic hypertension. Stroke. 1995 Aug;26(8):1319-24. doi: 10.1161/01.str.26.8.1319. PMID 7631329
- [Background] Sutton-Tyrrell K, Wolfson SK Jr, Kuller LH. Blood pressure treatment slows the progression of carotid stenosis in patients with isolated systolic hypertension. Stroke. 1994 Jan;25(1):44-50. doi: 10.1161/01.str.25.1.44. PMID 8266382
- [Background] Sutton-Tyrrell K, Alcorn HG, Wolfson SK Jr, Kelsey SF, Kuller LH. Predictors of carotid stenosis in older adults with and without isolated systolic hypertension. Stroke. 1993 Mar;24(3):355-61. doi: 10.1161/01.str.24.3.355. PMID 8446969
- [Background] Zeigler-Johnson CM, Holmes JL, Lassila HC, Sutton-Tyrrell K, Kuller LH. Subclinical atherosclerosis in relation to hysterectomy status in black women. Stroke. 1998 Apr;29(4):759-64. doi: 10.1161/01.str.29.4.759. PMID 9550508
- [Background] Franklin SS, Sutton-Tyrrell K, Belle SH, Weber MA, Kuller LH. The importance of pulsatile components of hypertension in predicting carotid stenosis in older adults. J Hypertens. 1997 Oct;15(10):1143-50. doi: 10.1097/00004872-199715100-00012. PMID 9350588
- [Background] Sutton-Tyrrell K, Bostom A, Selhub J, Zeigler-Johnson C. High homocysteine levels are independently related to isolated systolic hypertension in older adults. Circulation. 1997 Sep 16;96(6):1745-9. doi: 10.1161/01.cir.96.6.1745. PMID 9323056
- [Background] Lassila HC, Sutton-Tyrrell K, Schwartz F, et al: Antihypertensive Medication Use 5 Years Following the Systolic Hypertension in the Elderly Program. CVD Prevention, 3:229-234, 2000.
- [Background] Evans RW, Sankey SS, Hauth BA, Sutton-Tyrrell K, Kamboh MI, Kuller LH. Effect of sample storage on quantitation of lipoprotein(a) by an enzyme-linked immunosorbent assay. Lipids. 1996 Nov;31(11):1197-203. doi: 10.1007/BF02524295. PMID 8934453
- [Background] Sutton-Tyrrell K, Wildman R, Newman A, Kuller LH. Extent of cardiovascular risk reduction associated with treatment of isolated systolic hypertension. Arch Intern Med. 2003 Dec 8-22;163(22):2728-31. doi: 10.1001/archinte.163.22.2728. PMID 14662626